CLINICAL TRIAL: NCT04478162
Title: Investigation of the Effect of Family Integrated Care Method on Preparedness for Discharge
Brief Title: The Effect of Family Integrated Care on Preparing Parents With Premature Infants Hospitalized in the Neonatal Intensive Care Unit for Discharge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, öznur tiryaki, Nursing, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 16214662/050.01.04/14
Record Dates: First submitted 2020-06-27; First posted 2020-07-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Neonatal Intensive Care Unit; Parents
Keywords: premature; Family Integrated Care; discharge; readiness; parents
MeSH Terms: conditions — Premature Birth | interventions — Drainage

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: The randomization will be done through the program with the Uniform Resource Locator (URL) address httpp://www.randomizer.org and it is planned to work with 1 month intervention and 1 month control group to prevent the groups from being affected by each other.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): All phases of the FICare model have been implemented. Parents in the intervention group were included in a one-week training program within the scope of the Family Integrated Care model. A maximum of four couples attended the training in each session. A training program was also organized at weekend for those who could not attend it during the week. Training subjects consisted of the importance of breast milk, breastfeeding positions, hygienic care practices (eyes, nose, mouth, ears, skin, diaper change), bathing, nail clipping, kangaroo care, drug administration, first and emergency support, safe sleep, doctor check-up times, and vaccine follow-ups. Care practices were first shown on the model infant, and parents were asked to practice on the model. When the clinical stabilization of their infants was achieved, parents were asked to attend at least three caregiving sessions and stay in the hospital for an average of six to eight hours.
  Interventions: Other: Supporting parents who have premature babies to be ready for discharge with the training given within the scope of FICare model.
- Control Groups (No Intervention): Individuals received usual care provided by nurses from the time the premature infant was admitted to the NICU until discharge. The usual care process is carried on between the nurse and the mother. Mothers are allowed to perform limited care practices (bottom cleaning, breastfeeding) that the nurse considers appropriate. Mothers of babies who are planned to be discharged start staying in the hospital approximately 2 days before. Fathers are not included in the care and process. They are not allowed to stay in the hospital. Fathers are only informed and not included in the care.

INTERVENTIONS:
Other: Supporting parents who have premature babies to be ready for discharge with the training given within the scope of FICare model. — At least 1 week of FICare training for parents At least 4 hours of training on FICare for health professionals Trainings will be held between 13:30 and 15:30 in a training room with heat, light and seating arrangement (for parents who are not able to participate in the training during the week, trainings will be held at the appropriate time interval on the weekend .) Premature baby dummy on oral care, eye care, nose care, ear care, skin care, bath, attired in clothes,/removal, safe sleeping baby, safe transport, kangaroo care (physical contact), non-invasive drug application will be shown and the parents also will be asked to implement,
  Arms: Experimental

SUMMARY:
Physiological and structural features of premature infants differ from mature newborns. Families worry about touching their very sensitive and fragile babies, which are quite different from their expectations, and they seriously concern about how they will take care of their babies who are cared for by the specialist staff at the hospital when they are discharged to home. Different approaches and models are applied in the Neonatal Intensive Care Units (NICU) to prepare families, especially mothers, for the discharge process and to overcome these fears of the parents. However, most of the time, investigators observe in both researches and units that these approaches are not efficient. In this study, which investigators started with the questions as "What can investigators do better in this issue?" and "How can investigators help families more in this process?", investigator have seen that Family Integrated Care (FICare) model is applied in some clinics abroad and successful results have been obtained. However, investigators did not come across a study that applied this model and examined the effect of it on parents on being ready for discharge. Since this study will be a first in terms of both this aspect and the application of this model in our country, in this unique study, investigators aim to draw attention to this approach in our country, also contribute to keeping the premature babies healthy.

Research Hypotheses:

H0 There is no difference between the readiness for discharge of mothers and fathers included in the FICare model compared to the control group.

H1 The hypothesis of this study is that the mothers included in the FICare model have higher levels of discharge readiness than the control group.

H2 The hypothesis of this study is that the fathers included in the FICare model have higher levels of discharge readiness than the control group.

DETAILED DESCRIPTION:
Background: The Family Integrated Care (FICare) model is a modern approach that supports the participation of parents (excluding ventilation, monitor adjustments, vascular fluid and drug administration) developed in collaboration between parents and healthcare professionals, which is carried out gradually in the NICU (1). Parents are informed about the general development of the baby, brain and sensory development, motor and behavior development, care of the premature. In addition, parents are informed about what they can do about general body cleaning and care, especially in touch, attachment, skin-to-skin contact, breastfeeding and increased breast milk and diaper change (2).FICare; It is a care model with a 25% increase in the weight gain of premature babies, a 80% increase in breastfeeding rate, a 25% decrease in parental stress, a significant decrease in critical incident reports such as hospital infection and sudden infant death (3). The care that these babies receive in their first hours, days, weeks and months is vital to determine their future health and long-term outcomes. Evidence suggests that if parents are supported and encouraged to take care of their babies while in hospital, this will have better outcomes for both the baby and their family. FICare support not only reduces the length of hospital stay of parents, but also reduces the rate of re-hospitalization, and strengthens the bond between parents and babies. It helps parents feel safer when taking care of their babies, both in the hospital and at home (4).

A standard care model for discharge preparation is not applied to parents who have a premature baby in their NICU. Institutions make the decision to discharge with the opinions of the doctor and nurse working in the unit. With the FICare model, it is thought that parents will be prepared for discharge, bonding between parents and babies, fulfilling their parental roles, supporting babies' breastfeeding, reducing hospital stay, enhancing parental-employee communication, and increasing the quality of care services..

Premature infants who were hospitalized for at least seven days between February 6, 2020, and August 15, 2021, in the NICU of a training and research hospital formed the population of the study. In the study, the total number of parents was determined as 68 when the margin of error was 5%, the power level was 81.17%, and the effect size value was 0.70. At the end of the study, a post hoc power analysis was conducted to determine the adequacy of the sample size. As a result of the power analysis, for the details of the difference between the groups in terms of the scale score of fathers with premature babies in the neonatal intensive care unit, type 1 error: 0.05, n: 68 people, effect size = 1.990, and the power level according to the structure was determined as 1.000. To determine the difference in terms of the scale score of mothers with premature babies in the neonatal intensive care unit, type 1 error: 0.05, n: 68 people, effect size = 2.586 and power level according to temperature was determined as 1.000. These values show that the sample size is sufficient.

ELIGIBILITY:
Inclusion Criteria:

1. Birth of the infant at the 28th-34th weeks of gestation,
2. First parenting experience of the mother and the father,
3. Parents' willingness to participate in the study and being open to communication,
4. Mother having breast milk,
5. Participation of parents in the discharge training program.

Exclusion Criteria:

1. Undergoing a surgical intervention,
2. Death of the baby
3. Transfer of the baby to another hospital,
4. Failure of the parent to complete all phases of the study.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Parents with premature babies at NICU
Enrollment: 68 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
Family Integrated Care model and evaluation of routine care practicesevaluation) will increase the readiness of parents. | up to nine months
  With the questionnaire to be used separately for mothers (Preparedness for Discharge Scale of the Mother with a Premature Baby in the Neonatal Intensive Care Unit) and fathers (Preparedness for Discharge Scale of the Father with a Premature Baby in the Neonatal Intensive Care Unit) with premature babies, their readiness for discharge will be measured. A minimum score of 22, a maximum of 154 points are obtained from the form applied to mothers, a minimum of 20 and a maximum of 140 points from the form applied to fathers. High scores indicate that parents are ready for discharge.

SECONDARY OUTCOMES:
Premature infants weight (kg) | up to nine months
  Body weight will be measured every day from the day the baby is admitted to NICU until the day she is discharged.Body weight will be measured every day from the day the baby is admitted to NICU until the day she is discharged.
  Measurements obtained by the percentile curve are evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Nursan ÇINAR, Proffesor, Principal Investigator — Sakarya University
Locations (1):
- Sakarya Education and Training Hospital, Sakarya, Adapazarı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
* Planning of the study, literature review, development of data collection tools, preparation of training slides and videos, provision of materials to be used in the study (2 months)
  * Application of Family Integrated Care model, Collection of Data (10 months)
  * Statistical analysis and evaluation of results (1 months)
  * Writing the research report (2 months)

REFERENCES:
- [Derived] Tiryaki O, Cinar N, Caner I. The effect of family integrated care on preparing parents with premature infants hospitalized in the neonatal intensive care unit for discharge. J Perinatol. 2024 Jul;44(7):1014-1021. doi: 10.1038/s41372-024-01931-5. Epub 2024 Mar 18. PMID 38499753
- See also: httpp — https://pubmed.ncbi.nlm.nih.gov/31502862/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31502862/